CLINICAL TRIAL: NCT05113108
Title: Transcranial Ultrasound Screening of Nursery Unit Neonatesfor Brain Abnormalities in Assuit University Hospital
Brief Title: Transcranial Ultrasound Screening of Nursery Unit Neonatesfor Brain Abnormalities
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Basma Fawzy Abd Elhameed Ali (Other)
Responsible Party: Sponsor-Investigator, Basma Fawzy Abd Elhameed Ali, Resident Doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Neonatal cranial Ultrasound
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Brain Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CUS — All neonates undergoing CUS at nursery unit at assiut university hospital. Cranial ultrasound is performed with basic grayscale imaging. For optimal resolution and good overview, a multifrequency (5-10 MHz) linear or convex sector transducer is used. Imaging is obtained through the anterior fontanel in the coronal and sagittal planes.{12,13} Typically, six to eight coronal images are obtained beginning at the frontal lobes just anterior to the frontal horns and extending to the occipital lobes posterior to the lateral ventricle trigones.{14} The transducer is then rotated 90°, and approximately five images are obtained, including a midline sagittal view of the corpus callosum and cerebellar vermis in addition to bilateral parasagittal images beginning in the midline and progressing laterally through the peripheral cortex.Doppler ultrasound may be added to assess ischemic areas.{13-15}

SUMMARY:
* To investigate the prevalence of cerebral abnormal findings in neonates admitted at nursery unit.{11}
* to identify the associated clinical features and to better target neonatal CUS investigations.{11}

DETAILED DESCRIPTION:
Preterm birth is associated with various brain injuries. The earlier the period of gestation, more is the incidence of brain injuries. Brain injuries are known to be one of the most important factors leading to significant morbidity and mortality in these vulnerable preterm babies.{1} Cranial ultrasound (CUS) examinations have been performed on preterm infants to diagnose various perinatal brain injuries and for the prediction of long term outcomes.{2} Cranial ultrasonography (CUS) is the preferred modality to image the neonatal brain.{3} The advantages of CUS are numerous: it can be performed at the bedside with little disturbance to the infant, it is relatively safe, and can be repeated whenever needed, enabling visualization of ongoing brain maturation and the evolution of lesions.{4,5}

ELIGIBILITY:
Inclusion Criteria:

* All neonates suspected clinically to be suffered from brain lesions at nursery unit at assiut university hospitals

Exclusion Criteria:

* Patients above the age of 28 days

Ages: 1 Day to 28 Days | Sex: All
Age Groups: Child
Study Population: Neonates undergoing CUS at nursery unit at university hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Investigate the preavalence of cerebral abnormal findings in neonates | Baseline
  Cranial Ultrasound is performed with basic grayscale imaging

REFERENCES:
- [Background] Maalouf EF, Duggan PJ, Counsell SJ, Rutherford MA, Cowan F, Azzopardi D, Edwards AD. Comparison of findings on cranial ultrasound and magnetic resonance imaging in preterm infants. Pediatrics. 2001 Apr;107(4):719-27. doi: 10.1542/peds.107.4.719. PMID 11335750